CLINICAL TRIAL: NCT02082561
Title: False Safety Behavior Elimination Therapy: A Randomized Study of a Brief Individual Transdiagnostic Treatment for Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Florida State University
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Panic Disorder; Generalized Anxiety Disorder; Social Anxiety Disorder
Keywords: transdiagnostic treatment; cognitive behavior therapy; anxiety; panic disorder; generalized anxiety disorder; social anxiety disorder
MeSH Terms: conditions — Panic Disorder; Generalized Anxiety Disorder; Phobia, Social; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transdiagnostic Treatment (F-SET) (Experimental): F-SET treatment consisted of five weekly individual sessions (approximately 50 minutes each). The F-SET protocol is consistent with current CBT protocols for anxiety disorders.
  Interventions: Behavioral: Transdiagnostic Treatment (F-SET)
- Waitlist (No Intervention): The waitlist control condition was comprised of patients randomly assigned to the waitlist condition (WL). Individuals in this condition were reassessed after five weeks and were then offered treatment, but were no longer followed.

INTERVENTIONS:
Behavioral: Transdiagnostic Treatment (F-SET) — F-SET treatment consisted of five weekly individual sessions (approximately 50 minutes each). The participants learn to techniques and skills to help them reduce their anxiety. F-SET protocol is consistent with current CBT protocols for anxiety disorders.
  Arms: Transdiagnostic Treatment (F-SET)

SUMMARY:
The aim of the current study was to test the efficacy of an individually administered, brief (5-session) transdiagnostic treatment for anxiety disorders. The current treatment (called F-SET) focuses chiefly on the elimination of anxiety maintaining behaviors and cognitive strategies (so-called "safety" aids) among individuals suffering from a range of anxiety disorders including generalized anxiety disorder (GAD), social anxiety disorder (SAD) and panic disorder (PD). We hypothesized that the F-SET protocol would produce better overall outcome relative to a waitlist control.

DETAILED DESCRIPTION:
The aim of the current study was to test the efficacy of an individually administered, brief (5-session) transdiagnostic treatment for anxiety disorders. The current treatment (called F-SET) focuses chiefly on the elimination of anxiety maintaining behaviors and cognitive strategies (so-called "safety" aids) among individuals suffering from a range of anxiety disorders including generalized anxiety disorder (GAD), social anxiety disorder (SAD) and panic disorder (PD).

Four primary hypotheses were evaluated in the current study: (1) the F-SET protocol would produce better overall outcome relative to a waitlist control, (2) the F-SET protocol would yield clinically significant improvement of primary diagnosis symptoms as well as secondary diagnosis symptoms, (3) the F-SET protocol would create treatment improvement that is maintained during a 1 month follow-up interval and (4) given that reduction of safety aid use is the key mechanism of change in the F-SET treatment, a reduction in safety aid use will mediate the relationship between pre and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a primary diagnosis of panic disorder, generalized anxiety disorder, or social anxiety disorder.
* No change in medication type or dose during the 12 weeks prior to treatment

Exclusion Criteria:

* Current or past schizophrenia, bipolar disorder, or organic mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The Structured Clinical Interview for the DSM-IV | One Month Follow-up
  Structured Clinical Interview for the DSM-IV (SCID-IV). The SCID-IV (Spitzer, Gibbon, & Williams, 1996) is a structured diagnostic interview designed to provide detailed coverage of Axis-I disorders. The SCID-IV has been shown to be a reliable and valid measure of the Diagnostic and Statistical Manual of Mental Disorders (fourth edition-text revision; American Psychiatric Association, 2000) Axis I disorders (Zanarini et al., 2000).
Clinician Global Impressions Scale (CGI) - Severity of Illness Subscale | One Month Follow-up
  Clinician Global Impressions Scale (CGI) - Severity of Illness Subscale. The CGI (Guy, 1976) is a widely used clinician-rated measure of global impressions. The severity of illness subscale from the CGI is composed of a 7-point scale (ranging from 0=not at all ill to 6=among the most extremely ill patients) and is used to assess
Work and Social Adjustment Scale (WSAS) | One Month Follow-up
  Work and Social Adjustment Scale (WSAS). The WSAS is a 5-item descriptive measure of subjective interference in various life domains (i.e., work, home management, private leisure, and family relationships). Interference in the past week is rated from 0 (not at all interfering) to 8 (severe interference). The WSAS has demonstrated good internal consistency and has been successfully used in previous studies (e.g., Brown & Barlow, 1995; Ellard, Fairholme, Boisseau, Farchione, & Barlow, 2010). The WSAS was used as an index of overall disability and impairment. The WSAS demonstrated good internal consistency in the present sample (mean inter-item correlation = .28).

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Schmidt, Ph.D, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States